CLINICAL TRIAL: NCT02855424
Title: The Effect of Leg Cycling Exercise Program at Low or Moderate Intensity for Individuals With Subacute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KUMHIRB-F(II)-2016002
Record Dates: First submitted 2016-07-06; First posted 2016-08-04 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-06

CONDITIONS: Stroke
Keywords: stroke; exercise capacity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention): traditional rehabilitation merely, no ergocycling training
- the low-intensity exercise group (Experimental): traditional rehabilitation plus the low-intensity ergocycling exercise training
  Interventions: Other: the low-intensity exercise group
- the moderate-intensity exercise group (Experimental): traditional rehabilitation plus the moderate-intensity ergocycling exercise training
  Interventions: Other: the moderate-intensity exercise group

INTERVENTIONS:
Other: the low-intensity exercise group — Totally 20-time training, frequency 2-6 time/week, total 20 times.
  Arms: the low-intensity exercise group
Other: the moderate-intensity exercise group — Totally 20-time training, frequency 2-6 time/week,total 20 times.
  Arms: the moderate-intensity exercise group

SUMMARY:
Poor cardiopulmonary endurance is observed in individuals with acute stroke, even in chronic. In addition, the poor fitness may obstacle activities of daily life, decrease activities of autonomic system, and increase risks of recurrent, therefore, the cardiopulmonary endurance training should be included into the early-stage rehabilitation program. The ergocycling training could improve cardiopulmonary endurance for individuals with stroke. Moreover, the low-intensity exercise training can increase the willingness, and it is safer than the moderate-intensity exercise training. However, it needs to be evaluated whether the low-intensity exercise training can bring sufficient benefits, compared to the moderate-intensity exercise training. Objectives of the study is to compare the exercise benefits between the low-intensity and moderate-intensity exercise training, and then these would offer optimal exercise prescription and considerations in clinical practice.

DETAILED DESCRIPTION:
After giving their signed consent, subjects would be randomly assigned into the control group (traditional rehabilitation), the low-intensity exercise group (traditional rehabilitation plus low-intensity exercise training), or the moderate-intensity exercise group (traditional rehabilitation plus the moderate-intensity exercise training). Frequency of the exercise training is 2-6 times/week, totally 20 times. In the symptom-limit exercise tolerance tests, subjects wear a gas-collecting mask and electrocardiogram, and pre-set graduated loading was offered by the bike. One therapists and one doctor would monitor the test. For resistance and time setting within each exercise training, it is customized by results of exercise tolerance tests in baseline and the allocation. Moreover, a therapist would stay with subject ,monitor the training, and measure the blood pressure before and after the training.

ELIGIBILITY:
Inclusion Criteria:

1. the first-ever stroke
2. period of ischemic stroke onset is longer than two weeks, and less than six months, and the doctors agree with exercise training
3. unilateral hemiplegia
4. no obvious deficits of cognition. Scores of three items in the National Institutes of Health Stroke Scale are zero
5. be willing to join this study and give their consent

Exclusion Criteria:

1. aphasia
2. orthopedic problems (severe arthritis), neurologic injury (eg. peripheral nerve injury) that can interfere with movement of the lower limb, or cannot sit independently
3. with pace maker, severe cardiac arrhythmia, or heart failure
4. abnormal electrocardiography in rest, is not suitable for exercise tolerance test according to the American College of Sports Medicine guidance, for example, the atrioventricular block (AV block).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
changed value of symptom-limit exercise tolerance tests | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  One doctor and one therapist monitor the test. EKG and self-report are used.

SECONDARY OUTCOMES:
changed activity of autonomic nervous system (ANS) | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  The frequency domain analysis (measure unit of activity of ANS) is used in two conditions (sit and calculate math; 5 minutes/each condition).
10-meter walking test | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  Time of performing the 10 meters is measured.
changed score of the Barthel index | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  Using Barthel index questionnaire
changed score of the Stroke-Specific Quality of Life Scale (SSQOL) | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  Using SSQOL questionnaire
changed value of the Fugl-Meyer Assessment Lower Extremity (FMA-LE) | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  Measure items of FMA-LE
changed score of Multi-dimensional Fatigue Inventory | Baseline, 4 weeks to 10 weeks for exercise completion, one-month follow-up
  Using Multi-dimensional Fatigue Inventory questionnaire
performance of cycling | 4 weeks to 10 weeks for exercise completion
  the maximal power is recorded by a chip of the training bike continually during each training;2-6 times/week, total 20 times training.

CONTACTS AND LOCATIONS:
Overall Officials: Miao-Ju Hsu, PHD, Principal Investigator — Kaohsiung Medical University

IPD SHARING:
Plan to Share IPD: No